CLINICAL TRIAL: NCT05566366
Title: Understanding the Impact of Death Conditions Linked to the COVID-19 Health Crisis on the Grieving Process in Bereaved Families (Adolescents and Adults): a Qualitative Study
Brief Title: Understanding the Impact of Death Conditions Linked to the COVID-19 Crisis on the Grieving Process in Bereaved Families
Acronym: COVIDAAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP210638
Record Dates: First submitted 2022-06-27; First posted 2022-10-04 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Psychological Disorder
Keywords: COVID19 related psychological disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- population who lost a loved one during the COVID19 health crisis (Other): Analyze the grieving process of people who have lost a close first degree relative, understand the impact of death conditions on this process and model a "theory of mourning" in the context of the actual epidemic health crisis.
  Interventions: Other: Qualitative research interview

INTERVENTIONS:
Other: Qualitative research interview — Qualitative research interview Administration of quantitative scales

SUMMARY:
This study aims to analyze the grieving process of people who have lost a close first degree relative, understand the impact of death conditions and model a "theory of mourning" in the context of the COVID-19 crisis .

DETAILED DESCRIPTION:
The COVID-19 pandemic has confronted us with an unprecedented health crisis, this had major consequences on mental health . International literature has already shown an increase in psychological and psychiatric distress in patients followed in psychiatry, and in the general population.

For bereaved relatives, certain factors contribute to complicate the mourning process, such as: the absence of communication with the healthcare team, the prohibition of visits, the absence of funeral rites... In the proposed research, we will analyze the grieving process of people who have lost a close first degree relative in children and adolescents population, understand the repercussions conditions of death in bereaved families and model a "theory of mourning" in the context of the current epidemic health crisis.

ELIGIBILITY:
Inclusion Criteria:

* Bereaved person who lost a close relative (child, adolescent, adult) since March 2020
* Age over 15 years old
* First degree relative (husband-wife or equivalent, father-mother, son-daughter, brother-sister)
* A bereaved person who is in at least one of the following conditions:
* Unable to visit the hospital if hospitalized OR
* Unable to travel to the home/EPHAD/hospital OR
* Wish not to travel for personal reasons OR
* Failure to perform funeral rites OR
* Failure to respect the wishes of the deceased and his or her own wishes OR
* Inability to see the deceased OR
* Opportunity to participate in the funeral OR
* Unable to say goodbye OR
* Inability to communicate via telephone and/or smartphone OR
* Unable to repatriate the body to the country or region of origin
* Relative who died (child, adolescent, adult) between March 2020 and March 2021 with Covid-19 or other life-threatening conditions
* Relative who died in an inpatient or outpatient setting (EPHAD, home or other structure)
* French or non-French speaking bereaved person

Exclusion Criteria:

* Presence of a pathology preventing good elocution during the interview:

  * Presence of a neurological pathology (e.g. dementia, Alzheimer's, aphasia, dysphasia)
  * Presence of an unstabilised psychiatric disorder
* Person under guardianship or curatorship

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Identify the most traumatic aspects for bereaved families and better identify risk factors that may complicate the grieving process and contribute to the development of possible psychopathology. | 9 months
  In accordance with good practice in qualitative methodology, no secondary judging criteria should be used be provided

SECONDARY OUTCOMES:
Description of the socio-demographic characteristics of the bereaved | 9 months
  In accordance with good practice in qualitative methodology, no secondary judging criteria should be used be provided
Exploration of the relational aspects between the bereaved, his deceased and the rest of his family circle. | 9 months
  In accordance with good practice in qualitative methodology, no secondary judging criteria should be used be provided
Exploration of the history of the disease (Covid-19 and not Covid-19) and care management (extra-hospital and / or intra-hospital) until the announcement of the death | 9 months
  In accordance with good practice in qualitative methodology, no secondary judging criteria should be used be provided
Analysis of the relational dimensions between the bereaved and the healthcare team | 9 months
  In accordance with good practice in qualitative methodology, no secondary judging criteria should be used be provided
Exploration of support practices for the deceased (s) and funeral rites practices implemented by the bereaved | 9 months
  In accordance with good practice in qualitative methodology, no secondary judging criteria should be used be provided
Analysis of coping strategies and resilience factors of the bereaved person | 9 months
  In accordance with good practice in qualitative methodology, no secondary judging criteria should be used be provided
• Exploration of the dimensions of the lived experience and feelings of the grieving person • Exploration of the psychological state of the bereaved | 9 months
  In accordance with good practice in qualitative methodology, no secondary judging criteria should be used be provided
• Exploration of the bereaved person's experience of reporting the epidemic in the media and the COVID-19 disease (whether or not they have contracted it) | 9 months
  In accordance with good practice in qualitative methodology, no secondary judging criteria should be used be provided
• Assessment of pathological grief (Inventory of Complicated Grief - ICG) • Connor-Davidson ResilienceScale (CD-RISC) Resilience Assessment • Assessment of post-traumatic symptoms in adolescent Children'sRevised Impact of Events Scale (CRIES) | 9 months
  In accordance with good practice in qualitative methodology, no secondary judging criteria should be used be provided
Assessment of post-traumatic symptoms in adults (Post-Traumatic Stress Disorder) (Post-traumatic stress disorder checklist version DSM-5) (PCL-5) | 9 months
  In accordance with good practice in qualitative methodology, no secondary judging criteria should be used be provided
• Assessment of pathological grief (Inventory of Complicated Grief - ICG) | 9 months
  In accordance with good practice in qualitative methodology, no secondary judging criteria should be used be provided
Connor-Davidson ResilienceScale (CD-RISC) Resilience Assessment | 9 months
  In accordance with good practice in qualitative methodology, no secondary judging criteria should be used be provided
Assessment of post-traumatic symptoms in adolescent Children'sRevised Impact of Events Scale (CRIES) | 9 months
  In accordance with good practice in qualitative methodology, no secondary judging criteria should be used be provided
Hogan Inventory Bereavement - Short Form - Children and Adolescent Mourning Scale (HIB-SF-CA) | 9 months
  In accordance with good practice in qualitative methodology, no secondary judging criteria should be used be provided
Adolescent Resilience Assessment Child and YouthResilienceMeasure (CYRM-R) | 9 months
  In accordance with good practice in qualitative methodology, no secondary judging criteria should be used be provided

CONTACTS AND LOCATIONS:
Overall Officials: Carla DE STEFANO, Dr, Principal Investigator — Avicenne Hospital-APHP

REFERENCES:
- [Background] Xiong J, Lipsitz O, Nasri F, Lui LMW, Gill H, Phan L, Chen-Li D, Iacobucci M, Ho R, Majeed A, McIntyre RS. Impact of COVID-19 pandemic on mental health in the general population: A systematic review. J Affect Disord. 2020 Dec 1;277:55-64. doi: 10.1016/j.jad.2020.08.001. Epub 2020 Aug 8. PMID 32799105
- [Background] Shear MK, Ghesquiere A, Glickman K. Bereavement and complicated grief. Curr Psychiatry Rep. 2013 Nov;15(11):406. doi: 10.1007/s11920-013-0406-z. PMID 24068457
- [Background] Wallace CL, Wladkowski SP, Gibson A, White P. Grief During the COVID-19 Pandemic: Considerations for Palliative Care Providers. J Pain Symptom Manage. 2020 Jul;60(1):e70-e76. doi: 10.1016/j.jpainsymman.2020.04.012. Epub 2020 Apr 13. PMID 32298748
- [Background] Kersting A, Brahler E, Glaesmer H, Wagner B. Prevalence of complicated grief in a representative population-based sample. J Affect Disord. 2011 Jun;131(1-3):339-43. doi: 10.1016/j.jad.2010.11.032. Epub 2011 Jan 8. PMID 21216470
- [Background] Demartini B, Nistico V, D'Agostino A, Priori A, Gambini O. Early Psychiatric Impact of COVID-19 Pandemic on the General Population and Healthcare Workers in Italy: A Preliminary Study. Front Psychiatry. 2020 Dec 22;11:561345. doi: 10.3389/fpsyt.2020.561345. eCollection 2020. PMID 33414728
- [Background] Brooks SK, Webster RK, Smith LE, Woodland L, Wessely S, Greenberg N, Rubin GJ. The psychological impact of quarantine and how to reduce it: rapid review of the evidence. Lancet. 2020 Mar 14;395(10227):912-920. doi: 10.1016/S0140-6736(20)30460-8. Epub 2020 Feb 26. PMID 32112714